CLINICAL TRIAL: NCT05189860
Title: The C-MIC-II Follow-Up Study
Acronym: C-MIC-II-FU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berlin Heals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-MIC-II-FU
Record Dates: First submitted 2021-12-27; First posted 2022-01-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Systolic Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Study objective is to assess the safety of the C-MIC System in case of system extended use or abandonment or explantation in patients having received a C-MIC System in the context of a prior study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- C-MIC Device (Experimental): Device plus Standard of Care
  Interventions: Device: C-MIC system

INTERVENTIONS:
Device: C-MIC system — This study aims to follow up patients already treated with a C-MIC System over a period of 2 years following the initial treatment with the device, to assess the long term results.

SUMMARY:
The C-MIC System is a medical device used to treat heart failure per the intended purpose which is to treat heart failure by applying an electrical micro-current to the heart.

Target patients for this study are patients who have received the device in a prior study.

DETAILED DESCRIPTION:
The C-MIC System is a medical device used to treat heart failure per the intended purpose which is to treat heart failure by applying an electrical micro-current to the heart. The therapy with the C-MIC System is intended to take 6 months.

The C-MIC System consists of four parts, of which three are implanted: a transvenous and an epicardial lead and a power source to which the leads are connected. Both leads have the function to transmit micro-current to the heart. A Portable User Terminal (PUT) is needed for programming and readout of the data recorded by the Implantable Microcurrent Device (IMD).

Target patients of the C-MIC System at the time of implantation and inclusion in the C-MICII Study were patients with idiopathic dilative cardiomyopathy (NYHA class III - NYHA class who have systolic left ventricular dysfunction despite adequate therapy of heart failure.

Target patients for this study are patients who have received the device in a prior study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a C-MIC System during the C-MIC-II Study.
* Informed consent in writing from the patient.

Exclusion Criteria:

* Patients who are unwilling or unable to participate in the study visits.
* Vulnerable Patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  Rate of all cause, cardiac and device related mortality
Hospitalizations | 2 years
  Rate of all-cause, cardiac and device related hospitalizations
Adverse events | 2 years
  Overall incidence and severity of adverse events including malfunction

SECONDARY OUTCOMES:
Change in cardiac performance | 2 Years
  Left ventricular ejection fraction
Treatment adjustment | 2 Years
  Need for prolonged therapy with the C-MIC System in responder patients
Patient related outcome | 2 years
  Kansas City Cardiomyopathy Questionnaire (KCCQ: 0-100). Higher score represent better health status
Change in New York Heart Association (NYHA) classification | 2 years
  NYHA functional class
Cange in exercise ability | 2 years
  Cardiopulmonary exercise test
Change in aerobic capacity and endurance | 2 years
  6 Minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Peter Goettel, MD, Study Chair — Berlin Heals GmbH
Locations (6):
- Bosnia and Herzegovina (2):
  - University Clinical Centre of Republic of Srpska, Banja Luka, Banja Luka
  - University Clinical Center of Sarajevo, Sarajevo, Sarajevo
- Clinical Hospital Dubrava, Zagreb, City of Zagreb, Croatia
- University Clinic Cardiac Surgery, Skopje, North Macedonia
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Parent trial — https://clinicaltrials.gov/ct2/show/NCT04662034